CLINICAL TRIAL: NCT02761590
Title: Influence of a Circuit Trining Protocol on Intermuscular Adipose Tissue of Knee Osteoarthritis Patients: a Randomized Controlled Trial
Brief Title: Circuit Training on Knee Osteoarthritis Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidade Federal de Sao Carlos (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Principal Investigator, Aline Castilho de Almeida, MSc, Universidade Federal de Sao Carlos
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UFSCar - 2016
Record Dates: First submitted 2016-04-28; First posted 2016-05-04 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Knee Osteoarthritis
Keywords: intermuscular fat; circuit training; adipokines; inflammation; computed tomography scan
MeSH Terms: conditions — Osteoarthritis, Knee; Inflammation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Circuit training protocol (Experimental): The CT protocol will be held in three sessions per week for 14 weeks. The volume of work is defined by the training section of time and intensity of effort by the heart rate response to exercise.
  The construction of own model of periodization to be used complies with the biological principle of interdependence volume vs. intensity, and duration of 14 weeks, proposing a week of recuperative exercises after two weeks of stress, gradually increasing the intensity with respective volume settings. This model is based on the concepts described by Turner et al. that concludes in favor of the organization of training adapted to the reality of the public to be trained.
  Interventions: Other: Circuit training protocol
- Strength training protocol (Active Comparator): The strength training protocol was performed in three sessions per week for 14 weeks and divided into three levels.
  The initial load set for each exercise was based on the one repetition maximum test (1 RM). Strengthening exercises were performed in two sets of 15 repetitions, using 25% 1RM for hip adductors and abductors, and 50% 1RM for the quadriceps and hamstrings, using ankle weights. Exercises for the trunk were performed in 3 10-second series, increasing the duration when participants were able.
  Interventions: Other: Circuit training protocol
- Educational Protocol (No Intervention): In order to provide care, social interaction, and health education, an educational protocol was conducted. This protocol consisted in interactive presentations of 60 minutes, twice a month for 14 weeks, totaling 7 meetings. The topics addressed pathophysiology of osteoarthritis, and American College of Rheumatology (ACR) recommendations on nutrition, posture, and lifestyle.

INTERVENTIONS:
Other: Circuit training protocol — The construction of own model of periodization to be used complies with the biological principle of interdependence volume vs. intensity, and duration of 14 weeks, proposing a week of recuperative exercises after two weeks of stress, gradually increasing the intensity with respective volume settings. This model is based on the concepts described by Turner et al. which concludes in favor of the organization of training adapted to the reality of the public to be trained.
  Arms: Circuit training protocol; Strength training protocol

SUMMARY:
Introduction: The increase in intermuscular adipose tissue (IMAT) can contribute to muscle weakness and consequently on progression of knee OA. The prescription of exercise protocols has been used as a treatment strategy to minimize some of the bouts. Circuit training (CT) involves the combination of strength training and aerobic in the same session and has shown benefits in body composition and physical function. But the literature is unclear with respect to the influences of CT in the concentration of IMAT in the population with knee OA. Objective: To investigate the influence of a 14-week CT protocol in body composition and thigh IMAT concentration as well as cartilage degradation indicators and systemic inflammation and its impact on quality of life in patients with knee OA.

DETAILED DESCRIPTION:
This study presents a randomized controlled trial design. They will be selected 40 participants diagnosed with knee OA grades II and III, aged 40 and 65 years and BMI <30 kg / m2 were randomly divided into two groups: participants underwent training (trained group - TG) and not subjected to training ( untrained group - NTG). The participants trained group will undergo a periodized CT protocol of 14 weeks load progression, 3 times a week, with sessions last 15 minutes in the first weeks and will arrive 35 minutes in final weeks, and added 10 minutes between heating and cooling down. All subjects will conduct pre and post CT variables: IMAT thigh (computed tomography); body composition (Dual-energy X-ray absorptiometry - DXA), inflammatory biomarker concentrations: IL-1β, IL-6, IL-10, TNF-α, leptin and adiponectin and joint degradation biomarkers (uCTX-II and sCOMP), performance tests functional (six-minute walk, 30 seconds chair stand test and stair climb test), muscle strength (maximum voluntary isometric contraction - MVIC), WOMAC and KOOS questionnaires, and catastrophizing pain scale. During the training protocol, uCTX-II variables, sCOMP and MVIC will also be evaluated. To compare the groups will be applied the unpaired t-test. When found significant main effects, the Bonferroni test will be used to identify the statistically significant differences. To compare the collections times (pre, during and post TC) for uCTX-II variables, sCOMP and MVIC will be held repeated measures ANOVA with post hoc Bonferroni, and the WOMAC variables, KOOS, DXA, IMAT, functional testing and inflammatory cytokines (pre and post CT) will be held the paired t test. A significance level of 5% (p ≤ 0.05) will be adopted.

ELIGIBILITY:
Inclusion Criteria:

* aged between 40 and 65
* sedentary
* radiographically and clinically diagnosed with knee OA

Exclusion Criteria:

* performed physical therapy or exercise protocol up to 6 months prior to the beginning of the evaluations of this study
* previous knee surgeries
* previous history of trauma to the lower limb
* corticosteroid infiltration in knees in the 30 days prior to baseline
* prosthesis (partial or total) hip or knee arthritis
* use of chondroprotective
* cognitive deficits that compromise the understanding of tests and exercises
* body mass index (BMI) ≥30 kg / m²
* heart disease uncontrolled
* history of muscle injuries severe (above grade I)
* motor deficits due to neuromuscular disease
* cardiac pacemaker use
* chronic diseases
* impaired renal function, or any other medical condition that makes it impossible to participate in this study.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-03; Primary Completion 2018-12 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Change from baseline Intermuscular adipose tissue (IMAT) at 14 weeks | baseline and post intervention (week 14 - the analysis will be conducted on the first week immediately after the end of the training
  The concentration of intermuscular fat tissue will be measured by computed tomography. The images will be obtained through a CT scanner Multislice (Brilliance CT 16-slice, Phillips), located at the University Hospital of San Carlos. The examination will be conducted by experienced personnel under the supervision of a radiologist, developer of this study.
  The suggested protocol will provide an image related to the mid-thigh area of both legs. Quantification of intermuscular fat quadriceps muscle will be carried out by a slice thickness of 10 mm corresponding to half the distance between the greater trochanter and the intercondylar notch of the femur. The analyzes of the areas will be manually performed using the software OsiriX., And the area of interest selected by a scan, in accordance with the density of tissue decay rates for quantification of adipose tissue present in cm2.

SECONDARY OUTCOMES:
Body composition | baseline and post intervention (week 14 - the analysis will be conducted on the first week immediately after the end of the training
  For body composition analysis as it is used absorptiometry apparatus of X-ray Dual Energy (DXA, Hologic Discovery A, Benford, MA) using the three compartment model (lean mass, adipose tissue and body mineral density ), thus allowing to estimate the total body composition and body segment.
  The participant will be placed in the supine position and should remain without moving during the examination. To obtain better image, the subject should not use any type of metal, either as accessories or clothing. The results are transmitted to a connected to the machine computer and the examination of the report will provide data expressed in grams and percentage, are used to analyze data related to adipose tissue (g) Lean Mass (g) of the total composition (g) and percentage arms of adipose tissue (right and left), trunk and legs (right and left), gynoid regions and android beyond the total body composition.
Inflammation and degradation of cartilage biomarkers | baseline and post intervention (week 14 - the analysis will be conducted on the first week immediately after the end of the training
  Serum concentrations of IL-1-β, IL-6, TNF-α, IL-10, leptin, adiponectin and sCOMP will be measured by the ELISA (Enzyme-Linked Immuno Sorbent Assay) according to the manufacturers recommendations. Patients will be instructed to perform blood collection in the morning and remain at rest for 30 minutes before collection, especially for the evaluation of sCOMP. To assess the concentration of uCTX-II, participants will be instructed not to perform physical activities in a previous 24-hour period prior to collection, and collect urine in two specific containers (with a capacity of 80 ml each) a sample of the first urine day.
Muscle strength | baseline and post intervention (week 14 - the analysis will be conducted on the first week immediately after the end of the training
  The maximum voluntary isometric contraction (MVIC) extension and knee flexion will be measured using a dynamometer handheld (Lafayette Instruments, Lafayette, IN, USA). Previously the tests, familiarization will be performed. To evaluate the strength of the knee extensors, participants remain seated with angle of the hip in 90 ° of flexion and knee angle of 0 ° (full extension), not elastic bands being positioned on the hip to avoid compensation, and evaluation the knee flexors, participants will be asked to stay in the supine position, with hip and knee flexed to be tested at 90 °, legs and ankles relaxed on the bench, extended contralateral leg on the stretcher and arms extended beside the body.

OTHER OUTCOMES:
WOMAC questionaire | baseline and post intervention (week 14 - the analysis will be conducted on the first week immediately after the end of the training
  To assess pain, stiffness and physical function will use the questionnaire WOMAC (Western Ontario and McMaster Universities), a self-administered instrument that addresses the impact and restrictions specifically on the quality of life of patients with OA of the lower limbs. It is a questionnaire translated and validated for the Portuguese language. Composed of 24 reported auto issues, based on information in the 72 hours prior to their application, it is divided into three domains: pain, stiffness and physical function. Scoring is done using a Likert scale, wherein each question scored between 0 and 100, distributed as follows: 0 = none; 25 = little; Moderate = 50; = 75 intense and very intense = 100 59. The final score will be determined by the highest score in each area, causing pain, stiffness and physical function considered worse the higher the score achieved.
KOOS questionaire | baseline and post intervention (week 14 - the analysis will be conducted on the first week immediately after the end of the training
  The Knee injury and Osteoarthritis Outcome Score (KOOS) is a self reported specific joint measure developed to assess a broad spectrum of patients with knee injuries and OA, for pain and other symptoms, function in daily life, function in sports and recreation, and quality of knee-related life, being easy to use, evaluating the short- and long-term health problems related to the knee joint.
  The KOOS contains 42 items covering five subscales: pain, other symptoms, activities of daily living, sport and leisure activities and quality of life. A score of 0 (extreme problems) 100 (smoothly) can be obtained separately for each sub-range.
Catastrophizing Scale of Pain | baseline and post intervention (week 14 - the analysis will be conducted on the first week immediately after the end of the training
  The Pain Scale Catastrophizing it is a self-administered scale, easy and fast application, which allows the identification of individuals with psychological traits to catastrophizing. This instrument consists of 13 items, which the patient should report the degree of thought or feeling described with respect to pain, always respecting a degree of 5 points. The total score is given by the sum of all items, ranging from 0 to 52 points. It asked patients to answer the questions according to the thoughts and feelings that develop when affected by pain, regardless of the time of the interview the patient is in pain or not.
40 meters fasted paced walk test | baseline and post intervention (week 14 - the analysis will be conducted on the first week immediately after the end of the training
  Participants are invited to ride at high speed, but in the safest way possible by ume ditância 10 m, returning, and repitindo for a total distance of 40 m. The time for the test will be timed and will then be calculated execution speed of each participant.
30 seconds chair stand test | baseline and post intervention (week 14 - the analysis will be conducted on the first week immediately after the end of the training
  From the sitting position with your feet positioned in the same direction of the shoulders on the floor, arms crossed, the participant must raise completely the chair and then sit through back repeatedly for 30 seconds. The chair should be positioned against a wall. Should count the total number of the chair lift (up and sit is a repeat) per test. The same chair is needed for re-testing.
Stair climb test | baseline and post intervention (week 14 - the analysis will be conducted on the first week immediately after the end of the training
  Consist of up and down a flight of stairs with handrails, steps 12 and 16 cm. Participants should start standing task on a line with the hand placed on the railing. The command to start, should climb to the top of the stairs and immediately turn on and off using the same rail. The task should be performed as soon as possible. The total test time is timed (in seconds), whereas longer times indicate more committed physical function.

CONTACTS AND LOCATIONS:
Overall Officials: Aline C Almeida, MSc, Principal Investigator — Universidade Federal de Sao Carlos
Locations (1):
- Federal University of São Carlos, São Carlos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] de Almeida AC, Aily JB, Pedroso MG, Goncalves GH, Pastre CM, Mattiello SM. Reductions of cardiovascular and metabolic risk factors after a 14-week periodized training model in patients with knee osteoarthritis: a randomized controlled trial. Clin Rheumatol. 2021 Jan;40(1):303-314. doi: 10.1007/s10067-020-05213-1. Epub 2020 Jun 8. PMID 32514678
- [Derived] de Almeida AC, Aily JB, Pedroso MG, Goncalves GH, de Carvalho Felinto J, Ferrari RJ, Pastre CM, Mattiello SM. A periodized training attenuates thigh intermuscular fat and improves muscle quality in patients with knee osteoarthritis: results from a randomized controlled trial. Clin Rheumatol. 2020 Apr;39(4):1265-1275. doi: 10.1007/s10067-019-04892-9. Epub 2019 Dec 21. PMID 31865505
- [Derived] de Almeida AC, Pedroso MG, Aily JB, Goncalves GH, Pastre CM, Mattiello SM. Influence of a periodized circuit training protocol on intermuscular adipose tissue of patients with knee osteoarthritis: protocol for a randomized controlled trial. BMC Musculoskelet Disord. 2018 Nov 30;19(1):421. doi: 10.1186/s12891-018-2325-y. PMID 30497420